CLINICAL TRIAL: NCT00129233
Title: The Novel Antihypertensive Goal Of hYpertension With diAbetes - Hypertensive Events and ARb Treatment (NAGOYA-HEART) Study
Brief Title: Comparison of Valsartan With Amlodipine in Hypertensive Patients With Glucose Intolerance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nagoya University (Other)
Responsible Party: Principal Investigator, TOYOAKI MUROHARA, Proffesor, Nagoya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 169
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus
Keywords: cardiovascular disease; rennin-angiotensin system; calcium channel blocker; impaired glucose tolerance
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Glucose Intolerance | interventions — Valsartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valsartan (Active Comparator): Valsartan group treated with 80-160mg daily valsartan without Ca channel blockers or ACE inhibitors.
  Interventions: Drug: Valsartan
- Amlodipine (Active Comparator): Amlodipine group treated with 5-10mg daily amlodipine without ACE inhibitors or angiotensin receptor blockers.
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Valsartan — valsartan 80 to 160 mg daily
  Arms: Valsartan
Drug: Amlodipine — Amlodipine 5 to 10 mg daily.
  Arms: Amlodipine

SUMMARY:
Various guidelines recommended angiotensin converting enzyme (ACE) inhibitors or angiotensin Ⅱ receptor-1 blockers (ARBs) for hypertensive patients with diabetes on the basis of the cardiac- and reno-protective effects of these drugs. However, these recommendations could not be extrapolated to Japanese patients, because Japan has been known as a country with a low incidence of coronary artery disease and a high incidence of cerebrovascular disease. Furthermore, calcium channel blockers (CCBs) also were protective against renal function as well as ACE inhibitors in Japanese diabetic hypertensive patients. This study will test whether ARBs or CCBs are superior in treating Japanese diabetic hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension
* Clinical diagnosis of type 2 diabetes or impaired glucose tolerance

Exclusion Criteria:

* History of congestive heart failure, myocardial infarction, or coronary revascularization in the recent 6 months.
* Taking calcium channel blocker for the purpose of angina pectoris
* Reduced ejection fraction (< 40%)
* Second- or third-degree of atrioventricular block
* Severe hypertension (> 200/110 mmHg) or secondary hypertension
* History of stroke in the recent 6 months
* Serum creatinine > 2.5 mg/dl
* Estimated survival duration less than 3 years due to other conditions
* Pregnant woman or possibly pregnant woman

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2004-10; Primary Completion 2010-07 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Composite cardiovascular events including fatal or non-fatal myocardial infarction, fatal or non-fatal stroke, admission due to heart failure, coronary intervention and sudden cardiac death | At least 3 years of mean follow up period

SECONDARY OUTCOMES:
total death | At least 3 years of mean follow up period
cardiac function evaluated by ultrasonography | At least 3 years of mean follow up period
incidence of atrial fibrillation/flutter | At least 3 years of mean follow up period
control of blood glucose | At least 3 years of mean follow up period
renal function | At least 3 years of mean follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Toyoaki Murohara, MD, PhD, Principal Investigator — Department of Cardiology, Nagoya University Graduate School of Medicine
Locations (1):
- Department of Cardiology, Nagoya University Graduate School of Medicine, Nagoya, Aichi-ken, Japan

REFERENCES:
- [Background] Julius S, Kjeldsen SE, Weber M, Brunner HR, Ekman S, Hansson L, Hua T, Laragh J, McInnes GT, Mitchell L, Plat F, Schork A, Smith B, Zanchetti A; VALUE trial group. Outcomes in hypertensive patients at high cardiovascular risk treated with regimens based on valsartan or amlodipine: the VALUE randomised trial. Lancet. 2004 Jun 19;363(9426):2022-31. doi: 10.1016/S0140-6736(04)16451-9. PMID 15207952
- [Derived] Yamashita K, Kondo T, Muramatsu T, Matsushita K, Nagahiro T, Maeda K, Shintani S, Murohara T. Effects of valsartan versus amlodipine in diabetic hypertensive patients with or without previous cardiovascular disease. Am J Cardiol. 2013 Dec 1;112(11):1750-6. doi: 10.1016/j.amjcard.2013.07.043. Epub 2013 Sep 13. PMID 24035165
- [Derived] Muramatsu T, Matsushita K, Yamashita K, Kondo T, Maeda K, Shintani S, Ichimiya S, Ohno M, Sone T, Ikeda N, Watarai M, Murohara T; NAGOYA HEART Study Investigators. Comparison between valsartan and amlodipine regarding cardiovascular morbidity and mortality in hypertensive patients with glucose intolerance: NAGOYA HEART Study. Hypertension. 2012 Mar;59(3):580-6. doi: 10.1161/HYPERTENSIONAHA.111.184226. Epub 2012 Jan 9. PMID 22232134 (Retraction: PMID 30354774 Hypertension. 2018 Sep;72(3):e37-e38)
- [Derived] Matsushita K, Muramatsu T, Kondo T, Maeda K, Shintani S, Murohara T; NAGOYA HEART Study Group. Rationale and design of the NAGOYA HEART Study: comparison between valsartan and amlodipine regarding morbidity and mortality in patients with hypertension and glucose intolerance. J Cardiol. 2010 Jul;56(1):111-7. doi: 10.1016/j.jjcc.2010.03.004. Epub 2010 Apr 20. PMID 20409690